CLINICAL TRIAL: NCT06637605
Title: Clinical Evaluation of Different Restorative Materials in Deep Cavities
Brief Title: Clinical Comparison of Restorative Materials
Status: Active, not recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Muhammet Karadaş, Clinical Professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: RTEUDHFMKARADAS003
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries
Keywords: Dental caries; Restorative material; Composite resin; Deep caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Composite resin materials are the first treatment choice in direct restorations due to their good mechanical properties, excellent esthetic properties, conservative preparation, and successful clinical performance. However, resin-based composite materials in deep cavities are more likely to irritate the pulp tissue due to insufficient polymerization and residual monomer release. Therefore, glass ionomer-based restorative materials can be used more successfully in deep cavities. In addition, the hardening mechanisms of high-viscosity glass ionomer cement are the same as those of conventional glass ionomer cement, and their wear resistance, surface hardness, compression, and bending strength are increased. No clinical studies evaluate the performance of different restorative materials in deep cavities. This clinical study aims to evaluate the clinical performance of high-viscosity glass ionomer, bulk-fill composite, and conventional composite in deep cavities.

DETAILED DESCRIPTION:
This study was a double-blind (evaluator and patient) randomized controlled clinical study with three study groups with an equal allocation. Three different restorative materials were compared in deep cavities.

The treated patients were called back for controls after one week, six months, and twelve months. Restorations were evaluated clinically according to modified FDI criteria (marginal discoloration, color match, anatomical form, fracture and retention, marginal adaptation, contact point, post-operative sensitivity, secondary caries and periodontal response).

Clinical evaluation was performed by one qualified clinicians using a mirror and probe under reflector light. Bite-wing radiographs were taken from the patients who were called for controls at 6-moth and 12-month to evaluate the formation of secondary caries.

Differences between adhesives at each time period were evaluated using Fisher's Exact test. The effect of time on restorations was evaluated using Wilcoxon Signed rank test (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients aged 18 and over
* Patients with good oral hygiene.
* Vital teeth are to be included in the study.
* The presence of an antagonist and a contact tooth for the tooth to be restored.
* Teeth with deep caries lesions or radiographically reaching ¾ of the dentin but with a hard dentin region between the caries and the pulp according to ESE (European Society of Endodontology) criteria.

Exclusion Criteria:

* Patients with a history of bruxism and periodontal disease
* Patients under 18 years of age
* Spontaneous pain in the tooth to be restored
* Intense carious lesion reaching the entire thickness of the dentin according to ESE (European Society of Endodontology) criteria
* Observation of mechanical perforation during caries cleaning
* Patients suspected of pregnancy or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The characteristics of the teeth were recorded before the restorative procedures. Periapical radiographs were used to determine the status and extent of caries and any potential periodontal or periapical pathology that might require endodontic treatment. The treated teeth were vital, asymptomatic, and in occlusal contact. As a result of the clinical and radiographic evaluations, teeth with deep caries lesions according to the ESE (European Society of Endodontology) criteria or those with radiographically reaching ¾ of the dentin but with a hard dentin zone between the caries and the pulp were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
World Dental Federation criteria (FDI) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- 53020, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No